CLINICAL TRIAL: NCT00900133
Title: A Pilot Trial to Correlate Serum Levels of Calgranulin A and B With Estrogen Receptor Status Among Patients With Breast Cancer
Brief Title: Study of Calgranulin A/B Levels in Patients With Newly Diagnosed Stage I,II,III Breast Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Pink, PhD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE7104; P30CA043703 (NIH); CASE-7104 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood draw following diagnosis of breast cancer to assess levels of circulating tumor markers.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: immunoenzyme technique — Serum samples are evaluated by enzyme-linked immunosorbent assay for tumor marker expression.
Other: laboratory biomarker analysis — Blood draw following diagnosis of breast cancer to assess levels of circulating tumor markers, calgranulin A and calgranulin B.

SUMMARY:
RATIONALE: Measuring levels of calgranulin A and calgranulin B in the blood of patients with breast cancer in the laboratory may help doctors identify and learn more about biomarkers related to breast cancer.

PURPOSE: This laboratory study is measuring calgranulin A and calgranulin B levels in the blood of patients with newly diagnosed stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine circulating levels of calgranulin A and calgranulin B in patients with estrogen receptor negative or estrogen receptor positive, newly diagnosed, primary stage I-III adenocarcinoma of the breast.

OUTLINE: This is a pilot study.

Patients undergo a blood draw following diagnosis of breast cancer to assess levels of circulating tumor markers, calgranulin A and calgranulin B. Serum samples are evaluated by enzyme-linked immunosorbent assay for tumor marker expression.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the breast

  * Stage I-III disease
  * No evidence of metastatic disease
  * Newly diagnosed disease
* Hormone receptor status:

  * Estrogen receptor-positive- or -negative tumor

PATIENT CHARACTERISTICS:

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* No Crohn's disease
* No arthritis
* No psoriasis
* No lupus erythematosus
* No multiple sclerosis
* No other severe active inflammation
* Not C-reactive protein positive
* No HIV positivity
* No other serious medical or psychiatric illness

PRIOR CONCURRENT THERAPY:

Radiotherapy

* No prior radiotherapy for breast cancer

Surgery

* No prior organ transplantation

Other

* No prior systemic therapy for breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Newly Diagnosed Stage I,II,III Breast Cancer. Primary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Correlation between circulating levels of calgranulin A and calgranulin B and the presence of estrogen receptor negative breast cancer | upon diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: John Pink, PhD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States